CLINICAL TRIAL: NCT00613964
Title: The Effects of Carperitide on Short and Long-term Prognosis in Patients With Both Cardiac and Renal Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Nara Medical University (Other)
Responsible Party: Yoshihiko Saito, First Department of Internal Medicine, Nara medical university
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cardiol001
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2009-02

CONDITIONS: Heart Failure; Renal Failure
Keywords: Natriuretic Peptides; Heart Failure; Renal Failure
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Therapy (Placebo Comparator): Standard heart failure therapy excluding carperitide administration
  Interventions: Drug: Standard heart failure therapy
- Carperitide Therapy (Active Comparator): Addition of carperitide administration to standard heart failure therapy
  Interventions: Drug: Carperitide heart failure therapy

INTERVENTIONS:
Drug: Carperitide heart failure therapy — carperitide(alpha-human atrial natriuretic peptide, 0.025-0.05μg/kg/min)
  Other Names: Loop-diuretics etc + HANP
  Arms: Carperitide Therapy
Drug: Standard heart failure therapy — Loop diuretics, Aldosterone blockers, Beta blockers, ACE inhibitors, Angiotensin receptor blockers, Nitrates, digitalis
  Arms: Standard Therapy

SUMMARY:
Carperitide (alpha-human atrial natriuretic peptide) improves systemic hemodynamics in patients with heart failure through a vasodilatory action, a natriuretic action, and inhibition of the renin-angiotensin-aldosterone system and has been widely-used in Japan. However, a paucity of report is available on the effects of carperitide on short and long-term prognosis in patients with both cardiac and renal failure. The purpose of this study is to evaluate the effects of carperitide therapy on short and long-term prognosis in patients with both cardiac and renal failure, in comparison with standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure of any etiology, diagnosed according to Framingham criteria
* Estimated GFR </= 60 ml/min/1.73 m2)

Exclusion Criteria:

* Severe heart failure required percutaneous cardiopulmonary bypass support (PCPS)
* End-stage renal failure on maintenance dialysis
* Severe hepatic dysfunction
* Severe anemia
* Allergic history of carperitide
* Pregnant women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Unexpected rehospitalization for cardiovascular events, uremic symptom, initiation of maintenance dialysis, and kidney transplantation | at 6 months and 2 years

SECONDARY OUTCOMES:
All cause mortality | at discharge, 6 months, and 2 years
Sudden death | at discharge, 6 months, and 2 years
Cardiovascular death | at discharge, 6 months, and 2 years
Plasma B-type natriuretic peptide concentration | at discharge, 6 months, and 2 years
Estimated GFR | at discharge, 6 months, and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiko Saito, MD, PhD, Study Chair — First Department of Internal Medicine, Nara Medical University
Locations (1):
- First Department of Internal Medicine, Nara Medical University, Nara, Japan